CLINICAL TRIAL: NCT06730490
Title: Autonomic Nervous System Function in Hypoxic-Ischemic Infants Treated With Therapeutic Hypothermia
Brief Title: ANS Function in HIE Infants Treated With Therapeutic Hypothermia
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Guilherme Sant'Anna, MD, Associate Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: ANS STUDY 01
Record Dates: First submitted 2018-08-21; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: Autonomic Nervous System; Therapeutic Hypothermia; Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
After birth, babies that have suffered from oxygen deprivation may develop hypoxic-ischemic encephalopathy (HIE). Moderate or severe HIE has been associated with death or disability. Therefore, these infants are treated with therapeutic hypothermia (TH), which should be initiated within the first six hours of life. This study aims to investigate the autonomic nervous system (ANS) function of these infants. Thus far, no systematic evaluation of ANS function has been performed, despite its potential in providing important information. Current methods include clinical assessment of pupils size and reactivity, and measurements of heart/respiratory rates. Thus, ANS function evaluation is rather limited and prone to significant inter-examiner variability. This study propose a more comprehensive analysis of ANS function by investigating heart rate variability (HRV) and whole body skin temperature distribution, skin perfusion, axillary and esophageal temperature complexity. The investigators hypothesize that HRV analysis and a more thorough evaluation of ANS function could provide additional information associated with important clinical outcomes, which could eventually be tested clinically.

DETAILED DESCRIPTION:
1. Problem and Hypothesis:

   Globally, an estimated 1.8 to 7.7 infants per 1000 live term births suffer from perinatal asphyxia or oxygen deprivation. This remains an important cause of HIE. Seven randomized control trials have demonstrated that therapeutic hypothermia (TH) is a safe and effective therapy for infants with moderate and severe HIE if initiated within the first 6 h of life. TH increases the chances of survival without increasing the rates of neurodevelopmental disability.

   Investigations of these infants have focused mainly on daily neurological exams (modified Sarnat Score), electrical activity of the brain (amplitude integrated electroencephalography or aEEG and EEG), and brain imaging. No systematic evaluation of the ANS function has been performed despite its potential in providing important information. Current methods include clinical assessment of pupils size and reactivity, and measurements of heart/respiratory rates and are therefore limited and prone to significant inter-examiner variability. As such, in this study the investigators are planning to performing a more comprehensive analysis of ANS function under the hypothesis that in HIE infants treated with TH; a more thorough analysis of ANS function will provide additional information that can be associated with clinical outcomes.
2. Objectives:

   The objectives of the study are to measure and analyze the following variables of ANS function during TH and compare results between infants with and without poor outcomes:
   * Heart rate variability (primary outcome)
   * Skin temperature distribution and skin perfusion (secondary outcome)
   * Axillary temperature complexity (secondary outcome)
   * Esophageal temperature complexity (secondary outcome)

   A poor outcome will be defined as the composite of death, abnormal neurological exam at the end of the TH period or at discharge or transfer (whichever comes first), and abnormal brain MRI at day of life 10.
3. Methods and Analysis:

   For each newborn diagnosed with moderate or severe HIE and treated with TH, the investigators will collect demographics data using a pre-defined data collection form. Moreover, images of whole body temperature, recordings of axillary and esophageal temperature, and electrocardiogram (ECG), will be performed according to the following steps for days 1, 2 and 3 of TH:
   * Whole body infrared picture: infrared images (IR) of the whole infant will be obtained by using the E60bx camera (FLIR Systems, Inc. USA, Boston, MA). Whole body skin temperature will be analyzed by mapping temperature at the following areas: head, trunk, abdomen, upper and lower limbs, and upper and lower extremities. Mean ± SD and range values will be calculated for each area using the specific IR software. This will allow evaluation of skin temperature distribution for each patient for the specified study periods.
   * Skin perfusion: will be recorded by using the skin blood FlowMeter (ADInstruments, Bella Vista, Australia). A small surface probe will be placed at the abdomen just above the liver area using a self-adhesive ring.
   * Axillary temperature (Ta) and heart rate (HR): Ta will be recorded continuously for 1 h period using a probe placed at the R axilla and connected to the PowerLab data acquisition system®. The complexity of the temperature curve will be quantified using the approximate entropy (ApEn). HR will be measured by applying 3 ECG leads connected to a BioAmp and the PowerLab data acquisition system®. Heart rate variability (HRV) will be calculated using the time domain and frequency domain analysis, from 5 minutes segments of ECG and with the HRV module of the Labchart software®.
   * Esophageal temperature (Tes): will be collected every 5 minutes during the 1 h study period from the Blanketrol system device. Mean ± SD and the coefficient of variation of Tes values will be calculated.
4. Feasibility:

   Systematic evaluations of ANS function using the proposed study design and technologies have never been performed. Therefore, we will use a convenient sample size of 30 patients. In our NICU, approximately 40 infants with moderate and severe HIE are admitted and treated with TH every year. Thus, accounting for a 50-60% of loss to enroll due to refusal to consent, competing studies, unavailability of the research team, and patient instability, we estimate that we'll need a time frame between 24-30 months to achieve the calculated sample size of 30 patients. The same measurements will be performed in 15 patients with mild HIE (not cooled) as a control group.
5. Clinical Significance:

If any measurements of ANS function prove to be robust, they could have important implications for clinical practice. One aspect for future research is whether there is a correlation between ANS function and severity of disability or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Moderate or Severe HIE: 3 or more categories of the modified Sarnat Score in stage 2 or 3 (qualify for therapeutic hypothermia).
* Patients that are initiated on therapeutic hypothermia.
* Patients with Mild HIE, not treated with TH (control)

Exclusion Criteria:

-No encephalopathy, defined normal neurological exam.

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns admitted to the Montreal Children's Hospital neonatal intensive care unit (NICU) with mild, moderate or severe hypoxic-ischemic encephalopathy (HIE) and treated with therapeutic hypothermia (TH).
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | 6 months
  Heart rate variability (HRV) will be calculated using the time domain and frequency domain analysis and with the HRV module of the Labchart software®.

SECONDARY OUTCOMES:
Whole body skin temperature (WBST) | 6 months
  Whole body skin temperature (WBST): by using infrared (IR) images to map body temperature at the following areas: head, trunk, abdomen, upper and lower limbs, and upper and lower extremities. Mean ± SD and range values will be calculated for each area using the specific IR software.
Skin perfusion | 6 months
  Skin perfusion will be recorded by using the skin blood FlowMeter (ADInstruments, Bella Vista, Australia). A small surface probe will be placed at the abdomen just above the liver area using a self-adhesive ring.
Axillary temperature (Ta) | 6 months
  Axillary temperature (Ta) will be recorded continuously for 1 h period using a probe placed at the R axilla and connected to the PowerLab data acquisition system®.
Esophageal temperature (Tes) | 6 months
  Esophageal temperature (Tes): will be collected every 5 minutes during the 1 h study period from the Blanketrol system device. Mean ± SD and the coefficient of variation of Tes values will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme M Sant'Anna, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lawn J, Shibuya K, Stein C. No cry at birth: global estimates of intrapartum stillbirths and intrapartum-related neonatal deaths. Bull World Health Organ. 2005 Jun;83(6):409-17. Epub 2005 Jun 17. PMID 15976891
- [Background] Shankaran S, Laptook AR, Ehrenkranz RA, Tyson JE, McDonald SA, Donovan EF, Fanaroff AA, Poole WK, Wright LL, Higgins RD, Finer NN, Carlo WA, Duara S, Oh W, Cotten CM, Stevenson DK, Stoll BJ, Lemons JA, Guillet R, Jobe AH; National Institute of Child Health and Human Development Neonatal Research Network. Whole-body hypothermia for neonates with hypoxic-ischemic encephalopathy. N Engl J Med. 2005 Oct 13;353(15):1574-84. doi: 10.1056/NEJMcps050929. PMID 16221780
- [Background] Gluckman PD, Wyatt JS, Azzopardi D, Ballard R, Edwards AD, Ferriero DM, Polin RA, Robertson CM, Thoresen M, Whitelaw A, Gunn AJ. Selective head cooling with mild systemic hypothermia after neonatal encephalopathy: multicentre randomised trial. Lancet. 2005 Feb 19-25;365(9460):663-70. doi: 10.1016/S0140-6736(05)17946-X. PMID 15721471
- [Background] Zhou WH, Cheng GQ, Shao XM, Liu XZ, Shan RB, Zhuang DY, Zhou CL, Du LZ, Cao Y, Yang Q, Wang LS; China Study Group. Selective head cooling with mild systemic hypothermia after neonatal hypoxic-ischemic encephalopathy: a multicenter randomized controlled trial in China. J Pediatr. 2010 Sep;157(3):367-72, 372.e1-3. doi: 10.1016/j.jpeds.2010.03.030. Epub 2010 May 20. PMID 20488453
- [Background] Simbruner G, Mittal RA, Rohlmann F, Muche R; neo.nEURO.network Trial Participants. Systemic hypothermia after neonatal encephalopathy: outcomes of neo.nEURO.network RCT. Pediatrics. 2010 Oct;126(4):e771-8. doi: 10.1542/peds.2009-2441. Epub 2010 Sep 20. PMID 20855387
- [Background] Jacobs SE, Morley CJ, Inder TE, Stewart MJ, Smith KR, McNamara PJ, Wright IM, Kirpalani HM, Darlow BA, Doyle LW; Infant Cooling Evaluation Collaboration. Whole-body hypothermia for term and near-term newborns with hypoxic-ischemic encephalopathy: a randomized controlled trial. Arch Pediatr Adolesc Med. 2011 Aug;165(8):692-700. doi: 10.1001/archpediatrics.2011.43. Epub 2011 Apr 4. PMID 21464374
- [Background] Azzopardi DV, Strohm B, Edwards AD, Dyet L, Halliday HL, Juszczak E, Kapellou O, Levene M, Marlow N, Porter E, Thoresen M, Whitelaw A, Brocklehurst P; TOBY Study Group. Moderate hypothermia to treat perinatal asphyxial encephalopathy. N Engl J Med. 2009 Oct 1;361(14):1349-58. doi: 10.1056/NEJMoa0900854. PMID 19797281
- [Background] Laptook A, Tyson J, Shankaran S, McDonald S, Ehrenkranz R, Fanaroff A, Donovan E, Goldberg R, O'Shea TM, Higgins RD, Poole WK; National Institute of Child Health and Human Development Neonatal Research Network. Elevated temperature after hypoxic-ischemic encephalopathy: risk factor for adverse outcomes. Pediatrics. 2008 Sep;122(3):491-9. doi: 10.1542/peds.2007-1673. PMID 18762517
- [Background] Varela M, Churruca J, Gonzalez A, Martin A, Ode J, Galdos P. Temperature curve complexity predicts survival in critically ill patients. Am J Respir Crit Care Med. 2006 Aug 1;174(3):290-8. doi: 10.1164/rccm.200601-058OC. Epub 2006 May 11. PMID 16690981
- [Background] Varela M, Calvo M, Chana M, Gomez-Mestre I, Asensio R, Galdos P. Clinical implications of temperature curve complexity in critically ill patients. Crit Care Med. 2005 Dec;33(12):2764-71. doi: 10.1097/01.ccm.0000190157.64486.03. PMID 16352958
- [Background] Varela M, Jimenez L, Farina R. Complexity analysis of the temperature curve: new information from body temperature. Eur J Appl Physiol. 2003 May;89(3-4):230-7. doi: 10.1007/s00421-002-0790-2. Epub 2003 Mar 4. PMID 12736830
- [Background] Glass L. Synchronization and rhythmic processes in physiology. Nature. 2001 Mar 8;410(6825):277-84. doi: 10.1038/35065745. PMID 11258383
- [Background] Shankaran S, Laptook AR, Tyson JE, Ehrenkranz RA, Bann CM, Das A, Higgins RD, Bara R, Pappas A, McDonald SA, Goldberg RN, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Evolution of encephalopathy during whole body hypothermia for neonatal hypoxic-ischemic encephalopathy. J Pediatr. 2012 Apr;160(4):567-572.e3. doi: 10.1016/j.jpeds.2011.09.018. Epub 2011 Nov 1. PMID 22050871
- [Background] Rutherford M, Ramenghi LA, Edwards AD, Brocklehurst P, Halliday H, Levene M, Strohm B, Thoresen M, Whitelaw A, Azzopardi D. Assessment of brain tissue injury after moderate hypothermia in neonates with hypoxic-ischaemic encephalopathy: a nested substudy of a randomised controlled trial. Lancet Neurol. 2010 Jan;9(1):39-45. doi: 10.1016/S1474-4422(09)70295-9. Epub 2009 Nov 5. PMID 19896902